CLINICAL TRIAL: NCT04352231
Title: From Mouse to Man: Translating Findings in Mouse Study Into a Human Cohort (Luxembourgish Fiber Cohort: Lux-FiCo)
Brief Title: Luxembourgish Fiber Cohort
Acronym: Lux-FiCo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Centre Hospitalier du Luxembourg (Other); Integrated Biobank of Luxembourg (Other); University of Luxembourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LUX-FICO
Record Dates: First submitted 2020-02-26; First posted 2020-04-20 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Dietary Fiber; Gastrointestinal Microbiome; Healthy Volunteers
Keywords: Metagenome; Whole Genome Sequencing; Biomarkers; Mucolytic Activity; Mass cytometry; Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: This study involves recruitment of healthy volunteers to participate in a 2x2 crossover design controlled-diet study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High to Low Fiber Diet Intervention (Experimental): Participants receive the high fiber diet intervention first, then undergo a washout period to reverse any changes from the diet before receiving the low fiber diet intervention. A second washout period will follow this diet so that we can track any reversal of diet-linked changes.
  Interventions: Dietary Supplement: High Fiber Diet Intervention; Dietary Supplement: Low Fiber Diet Intervention
- Low to High Fiber Diet Intervention (Experimental): Participants receive the low fiber diet intervention first, then undergo a washout period to reverse any changes from the diet before receiving the high fiber diet intervention. A second washout period will follow this diet so that we can track any reversal of diet-linked changes.
  Interventions: Dietary Supplement: High Fiber Diet Intervention; Dietary Supplement: Low Fiber Diet Intervention

INTERVENTIONS:
Dietary Supplement: High Fiber Diet Intervention — Plant-based diet with a targeted quantity of 35 g of dietary fiber per day, from a variety of fiber types. Each meal will be balanced to provide all essential nutrients and portions will be of adequate size to ensure participants are satiated. Participants on both diet interventions will be given multivitamin supplements in order to ensure they are receiving essential vitamins and minerals.
Dietary Supplement: Low Fiber Diet Intervention — Animal based diet (meat, dairy) with a targeted quantity of 10 g of dietary fiber per day. Each meal will be balanced to provide all essential nutrients and portions will be of adequate size to ensure participants are satiated. Participants on both diet interventions will be given multivitamin supplements in order to ensure they are receiving essential vitamins and minerals.

SUMMARY:
Many human populations across the world are deficient in the intake of dietary fiber. This decline in fiber consumption parallels an increase in prevalence of a multitude of diseases (e.g. colorectal cancer, multiple sclerosis). A possible link for this association between dietary changes and the diseases could rest in the trillions of commensal gut microbes that digest dietary fibers, provide energy for colonic cells, and modulate the immune system. However, the molecular mechanisms that link fiber deficiency via the activities of the gut microbiome to various diseases have been poorly understood. The investigators previously showed that, in a mouse model with a defined human gut microbiota, removal of fiber from the diet favors proliferation of bacteria that degrade the gut's protective mucus lining. In the proposed project, the investigators aim to translate our findings from mouse studies to humans using a 2x2 crossover study among healthy adults. Forty participants will be randomly assigned to a low- or high-fiber dietary intervention and then, following a washout period to reverse any changes, switched to the other diet type. By employing longitudinal sampling of stool collections, the investigators envision that participants will exhibit increased abundance and activities of mucolytic bacteria when fed a low-fiber diet. The unique selling point of the proposed study involves setting up high-throughput culture collections of mucus-degrading bacteria, whose abundances and activities will be investigated by sequencing and enzymatic assays in stool. Additionally, the investigators will measure inflammatory markers in blood using CyTOF to assess whether short-term fiber deficiency exerts detectable changes in the host immune function. Thus, the proposed dietary intervention clinical trial will help elucidate the role of fiber deficiency in various chronic diseases.

DETAILED DESCRIPTION:
Industrialized nations tend to consume less dietary fiber and, in many nations with a Western-style diet, average consumption is half the recommended daily intake of 25-38 g/day. Dietary fiber is an important component of a healthy diet because it increases fecal bulking and laxation, lowers cholesterol and regulates levels of blood glucose. The connection between low fiber-intake and disease may rest with the gut microbiota, the trillions of commensal microorganisms that inhabit the gastrointestinal tract. Bacteria found in the gut are responsible for an array of functions that support human health, including conversion of host-indigestible fibers into short chain fatty acids (SCFAs), which provide energy for colonic cells, support mucus production, and modulate the immune system.

The investigators have recently investigated the effects of a fiber-free diet in a gnotobiotic mouse model with a 14-member synthetic microbial community showing that mucus-degrading bacteria outcompete fiber-degrading bacteria, causing degradation of the colonic mucus layer. One member of this synthetic community, Akkermansia muciniphila, is a commensal bacterium found at 1-4% relative abundance in the human gut and feeds specifically on the host-secreted mucins. However, this bacterium is significantly enriched in the gut of patients with multiple sclerosis and colorectal cancer, suggesting that its mucolytic capabilities may play a role in these diseases. A microbial shift toward enrichment of mucolytic bacteria could be an important precursor to gut-linked diseases. While observational studies have identified a lower risk of irritable bowel diseases (IBD) in people who consume diets high in fiber, fruits, and vegetables, no study has explicitly investigated the effects of fiber on the functional capacity of the human gut microbiome in the context of effects on the mucus-degrading microbiome. Based on our published work in mice, for the current project, the investigators hypothesize that deficiency of dietary fiber in humans promotes increased activities of mucus-degrading bacteria, thereby reducing the mucus lining in the intestine. The investigators request pump priming to initiate this pilot project, as it will generate foundational datasets to inform numerous follow-up studies.

Thus, the current project seeks to translate findings from mouse models to humans, using a crossover study among healthy adults. Participants will be randomly assigned to a first dietary intervention that is low or high in fiber and then, following a washout period intended to reverse any compositional changes, switched to the second diet type. The diets will be evaluated by a nutritionist to ensure that they differ in fiber content, but are comparable in terms of caloric and macronutrient content. The targeted amount of dietary fiber intake from the high-fiber test meals will be around 30 g/d more than the low-fiber diet. In addition to dietary records, the investigators will administer questionnaires, obtain basic clinical measures (blood pressure, weight, height, waist/thigh circumference), collect blood samples for immunological assays and collect stool samples before and at the end of each diet intervention for sequencing and functional profiling of bacterial communities.

The investigators will recruit healthy volunteers to participate in a 2x2 crossover design controlled-diet study. After statistical consultation, the investigators conclude that the investigators require a sample size of n=15 in each sequence group (a total sample size of N=30) to have 87.5% power to detect a -0.5 difference in means for alpha diversity (Shannon index) under the two diet conditions. Volunteers who meet all inclusion and exclusion criteria will be randomly assigned to a high- or low-fiber diet intervention and then, after a week-long washout period, will receive the second diet type. High and low fiber meals containing a variety of fiber types will be served to participants at a designated drop-off site (home or workplace) for one week in order to decrease variance in fiber intake, increase adherence to the diet, and maximize knowledge of the nutritional content in participants' diet. Nutritionally balanced dietary interventions are designed by a qualified dietitian at SERVIOR in conjunction with the LIH study team and delivered by Paul Eischen Traiteur, a partner catering service. Participants on both diet interventions will be given multivitamin supplements in order to further ensure they receive essential vitamins and minerals.

At the baseline visit, our team will work with nurses from the Clinical and Epidemiological Investigation Center (CIEC, headed by Dr. Manon Gantenbein) to collect demographic data, anthropometry, early life history, family medical history, detailed dietary patterns, and biological samples (blood, urine, and stool). Participants will use a Participant Diary to log their diet throughout the study in the form of daily 24 hour food recalls, except for foods or beverages provided during the dietary interventions. After each intervention period, a week-long washout period will be employed to reverse any changes that occurred due to the diet.

Mid-way through each intervention and washout period, the investigators will administer a brief survey containing questions relevant to our research objective. At each of these visits, CIEC nurses will collect biological samples and anthropometric measures. Participants will also be asked to drop off a stool sample for the next two days. All participant data will be pseudonymized when exported from Research Electronic Data Capture application (REDCap) for analysis and will be handled in accordance with the General Data Protection Regulation (GDPR). The study has been granted ethical approval by the Luxembourg Ministry of Health (Ref# 835x38895) and by Comité National d'Ethique de Recherche (CNER; Ref# 201911/03).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female:

   a. The investigators will aim for a 50:50 male:female ratio, at most 40:60. Therefore, given a sample size of N=40, if 24 eligible participants are exceed for one gender, the investigators will proceed with recruitment only for members of the underrepresented gender.
2. Between 18 and 35 years of age (expand to 55 if needed)
3. BMI between 18.5 ≥ BMI > 25 kg/m2 (expand to 30 if needed)
4. Born in Europe
5. Current resident of Luxembourg City or Esch-sur-Alzette (expand to nearby communes if needed)
6. Own a smartphone with access to Android or Apple Store applications

Exclusion Criteria:

1. Following a specific diet or subject to dietary restrictions for any reason
2. "Vigorous" physical activity level based on the International Physical Activity Questionnaire - Short Form (IPAQ-SF) criteria
3. Antibiotics usage within the past 3 months
4. Probiotics usage within the past 1 month
5. Laxatives usage within the past 1 month
6. Other regular medication usage (e.g. ibuprofen, warfarin)
7. Current or former smoker
8. Gastrointestinal disorder (e.g. ulcerative colitis, Crohn's disease) diagnosis
9. History of gastrointestinal surgery (excluding appendectomy)
10. Metabolic disorder diagnosis or predisposition (determined by blood test at eligibility screen)

    1. Prediabetes: fasting glucose 100-125 mg/dL (6.1-7.0 mmol/L) and/or drug treatment of elevated glucose (8)
    2. Diabetes: fasting glucose ≥126 mg/dL (7.0 mmol/L) and/or drug treatment of elevated glucose and/or previously diagnosed type 1 or type 2 diabetes (8)
    3. Hypertriglyceridaemia: fasting triglycerides ≥1.7 mmol/L (≥150 mg/dL) and/or drug treatment for elevated triglycerides (9)
    4. Hypercholesterolaemia: Fasting High-density lipoprotein cholesterol (HDL-C) < 40 mg/dL (< 1.0 mmol/L) in men and < 45 mg/dL (< 1.2mmol/L) in women and/or drug treatment for reduced HDL-C (9)
    5. Hypertension: Systolic BP ≥130 and/or diastolic BP ≥80 mm Hg and/or drug treatment of previously diagnosed hypertension (10)
11. Cancer (any type) diagnosis (note that a history of cancer that has been in remission for >3 years may still be considered eligible)
12. Immunodeficiency disorder (e.g. HIV) or autoimmune disorder (e.g. rheumatoid arthritis, lupus) diagnosis
13. Neurological disorder (e.g. advanced dementia, diagnosed major depressive disorder or generalized anxiety disorder)
14. Coagulation problems (e.g. hemophilia) or anemia impacting ability to participate in blood draw
15. Circulatory disorder (e.g. ischemic heart diseases or history of stroke)
16. Currently pregnant or lactating (breastfeeding)
17. Vacation planned during study period
18. Moving out of Luxembourg during the study period
19. Potential conflict of interest: involved in study design, administration, data analysis, or publication of findings or belonging to the lab group of the study's principal investigators

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Change in gut microbiota composition across study periods | through study completion, an average of 1 month
  Assessment of whether statistically significant shifts in the community composition has occurred will be performed using PERMANOVA on the SILVA-annotated taxonomic output of 16S rRNA gene sequence data from stool taken on the last three days of each intervention. Visual presentation of beta-diversity will be presented using PCoA plots based on weighted and unweighted Unifrac distance measures.

SECONDARY OUTCOMES:
Change in gut microbiota CAZyme abundance across study periods | through study completion, an average of 1 month
  Abundance of carbohydrate active enzymes (CAZymes) detected by shotgun sequencing of genomic DNA isolated from stool. Main comparison will be between high and low fiber diet intervention periods.
Change in gut microbiota mucolytic enzyme activity across study periods | through study completion, an average of 1 month
  Average bacterial sulfatase enzymatic activity of samples taken turing the last 3 days of each study period. Main comparison will be the average activity levels between high and low fiber diet intervention periods.

OTHER OUTCOMES:
Change in fecal acetate levels across study periods | through study completion, an average of 1 month
  Acetate concentrations by mass spectrophotometry over last 3 days of each study period.
Change in fecal propionate levels across study periods | through study completion, an average of 1 month
  Propionate concentrations by mass spectrophotometry over last 3 days of each study period.
Change in fecal butyrate levels across study periods | through study completion, an average of 1 month
  Butyrate concentrations by mass spectrophotometry over last 3 days of each study period.
Change in CyTOF immune profiles across study periods | through study completion, an average of 1 month
  Changes to the immune cell populations, profiled using Time of Flight Mass Cytometry (CyTOF).
Change in CRP across study periods | through study completion, an average of 1 month
  Changes to levels of C reactive protein (CRP), a general inflammatory marker, assayed using ELISA kits.
Change in LCN2 across study periods | through study completion, an average of 1 month
  Changes to levels of lipocalin-2 (LCN2), a general inflammatory marker, assayed using ELISA kits.
Change in calprotectin across study periods | through study completion, an average of 1 month
  Changes to levels of calprotectin, a general inflammatory marker, assayed using ELISA kits.
Change in fasting glucose level across study periods | through study completion, an average of 1 month
  Changes to levels of fasting glucose assayed by a commercial lab.

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh S Desai, PhD, Principal Investigator — Luxembourg Institute of Health
Locations (2):
- Luxembourg (2):
  - Luxembourg Institute of Health, Esch-sur-Alzette
  - Luxembourg Institute of Health, Strassen

IPD SHARING:
Plan to Share IPD: Yes
Sequencing data from microbiome samples and isolates will be uploaded to public repositories (ENA/EBI). Pseudonymized participant data will also be shared with collaborators and may be available to other researchers upon request and based on the participants sharing preferences as indicated in the consent form.
Time Frame: Data will become available to share with other researchers at the time of publication. Accession numbers for sequencing data will be published in the manuscript.
Access Criteria: All IPD will be pseudonymised. Researchers requesting use of this data should make an inquiry by email to the Principal Investigator explaining the purpose of their proposed work and what types of metadata they are interested in before any data sharing can be approved. In keeping with data minimization policies, we will share only the data that is relevant for the proposed analyses. Furthermore, data may not be shared if the participant has indicated on their consent form that they do not wish their data to be used in follow up studies (in the same or a different field of research).

REFERENCES:
- [Background] Martens EC, Neumann M, Desai MS. Interactions of commensal and pathogenic microorganisms with the intestinal mucosal barrier. Nat Rev Microbiol. 2018 Aug;16(8):457-470. doi: 10.1038/s41579-018-0036-x. PMID 29904082
- [Background] Desai MS, Seekatz AM, Koropatkin NM, Kamada N, Hickey CA, Wolter M, Pudlo NA, Kitamoto S, Terrapon N, Muller A, Young VB, Henrissat B, Wilmes P, Stappenbeck TS, Nunez G, Martens EC. A Dietary Fiber-Deprived Gut Microbiota Degrades the Colonic Mucus Barrier and Enhances Pathogen Susceptibility. Cell. 2016 Nov 17;167(5):1339-1353.e21. doi: 10.1016/j.cell.2016.10.043. PMID 27863247
- [Background] Belzer C, de Vos WM. Microbes inside--from diversity to function: the case of Akkermansia. ISME J. 2012 Aug;6(8):1449-58. doi: 10.1038/ismej.2012.6. Epub 2012 Mar 22. PMID 22437156
- [Background] Weir TL, Manter DK, Sheflin AM, Barnett BA, Heuberger AL, Ryan EP. Stool microbiome and metabolome differences between colorectal cancer patients and healthy adults. PLoS One. 2013 Aug 6;8(8):e70803. doi: 10.1371/journal.pone.0070803. Print 2013. PMID 23940645
- [Background] Jangi S, Gandhi R, Cox LM, Li N, von Glehn F, Yan R, Patel B, Mazzola MA, Liu S, Glanz BL, Cook S, Tankou S, Stuart F, Melo K, Nejad P, Smith K, Topcuolu BD, Holden J, Kivisakk P, Chitnis T, De Jager PL, Quintana FJ, Gerber GK, Bry L, Weiner HL. Alterations of the human gut microbiome in multiple sclerosis. Nat Commun. 2016 Jun 28;7:12015. doi: 10.1038/ncomms12015. PMID 27352007
- [Background] Hou JK, Abraham B, El-Serag H. Dietary intake and risk of developing inflammatory bowel disease: a systematic review of the literature. Am J Gastroenterol. 2011 Apr;106(4):563-73. doi: 10.1038/ajg.2011.44. PMID 21468064
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217